CLINICAL TRIAL: NCT05820516
Title: Cardiovascular, Renal and haemodynamIc Outcomes in Patients With Severe TrIcuspid Regurgitation After triCvALve System Implantation: an International Registry - CRITICAL INTERNATIONAL REGISTRY
Brief Title: Patients With Severe TrIcuspid Regurgitation After triCvALve System Implantation
Acronym: CRITICAL
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Marco De Carlo, M.D., Azienda Ospedaliero, Universitaria Pisana
Other Study IDs: CRITICAL
Record Dates: First submitted 2023-03-28; First posted 2023-04-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Severe Tricuspid Valve Regurgitation
Keywords: Severe Tricuspid Valve Regurgitation; TricValve
MeSH Terms: conditions — Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TricValve implantation — TricValve implantation

SUMMARY:
International Registry to collect patients with severe TR undergoing TricValve implantation from multiple Italian and European centers, aimed at:

* Assessing the effect of TricValve implantation on cardiovascular and all-cause mortality, HF rehospitalization, renal function, functional capacity and quality of life.
* Clarifying the haemodynamic effects of TricValve implantation and investigating their pathophysiological implications.

DETAILED DESCRIPTION:
Study Design

Type of study: Non-profit, multi-center, observational, prospective cohort study (with retrospective inclusion of the first cases performed)

Patient population: 100 patients

Date of beginning of enrollment: April 1st, 2023 (plus inclusion of patients treated since 2022)

Duration of the study: 12 months

All patients enrolled will undergo serial evaluations (Figure 1).

* At Baseline we will collect (see eCRF):

  * Clinical data regarding medical history, clinical status and medications;
  * Biohumoral data (blood and urine chemistry);
  * Haemodynamic data (Right Heart Catheterization);
  * Echocardiographic data including Comprehensive 2D and Doppler Transtoracic Echocardiography and Transoesophageal Echocardiography;
  * Anatomical data (Cardiac CT).
* At the time of procedure we will collect (see eCRF):

  * Procedural data including the occurrence of peri-procedural complications;
  * Haemodynamic data (Right Heart Catheterization).
* At discharge we will collect (see eCRF):

  * Clinical data regarding clinical status and medications;
  * Biohumoral data (blood and urine chemistry);
  * Echocardiographic data including comprehensive 2D and Doppler Transtoracic Echocardiography;
  * Peri-procedural data including the occurrence of peri-procedural complications.
* At 30-day follow-up we will collect (see eCRF):

  * Clinical data regarding medical history, clinical status and medications;
  * Biohumoral data (blood and urine chemistry);
  * Echocardiographic data including comprehensive 2D and Doppler Transtoracic Echocardiography;
* At 6-month follow-up we will collect (see eCRF):

  * Clinical data regarding medical history, clinical status and medications;
  * Biohumoral data (blood and urine chemistry);
  * Echocardiographic data including comprehensive 2D and Doppler transthoracic echocardiography;
  * Haemodynamic data (Right Heart Catheterization), if clinically indicated.
* At 1-year follow-up we will collect (see eCRF):

  * Clinical data regarding medical history, clinical status and medications;
  * Biohumoral data (blood and urine chemistry);
  * Echocardiographic data including Comprehensive 2D and Doppler Transtoracic Echocardiography;
  * Haemodynamic data (Right Heart Catheterization), if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18 years of age or older
2. The subject must be a patient with massive or torrential symptomatic tricuspid regurgitation demonstrated by echocardiography with significant backflow in the IVC and/or SVC and with a v-wave ≥ 25 mmHg as demonstrated by right heart catheterization (measured in the IVC and/or SVC 2-4 cm above/ below right atrium (RA) inflow) within 8 weeks prior to the implantation
3. Suitable for TricValve Transcatheter Bicaval Valves System implantation according to anatomic criteria by computed tomography (CT)
4. The subjects must have severe, tricuspid regurgitation leading to New York Heart Association (NYHA) class III or IV
5. Distance covered in 6-minute walk test (6MWT) ≥ 60m
6. Patient/authorized legal guardian understands the nature of the procedure, is willing to comply with associated follow-up evaluations, and provides written informed consent Patient/patient's authorized legal guardian is geographically stable (or willing to return for required study follow-up) and understands and is willing to fulfil all of the expected requirements of the clinical protocol

Exclusion Criteria:

1. Known significant intracardiac shunt (e.g. ventricular septal defect) or congenital structural heart disease based on heart team decision
2. Requirement for other elective cardiac procedures e.g. Percutaneous Coronary Intervention (PCI) or Coronary Artery Bypass Graft (CABG) up to 90 days after the procedure or 30 days before the procedure
3. Right ventricular failure (TAPSE ≤13 mm)
4. Systolic pulmonary arterial pressure > 65 mmHg as assessed by Doppler echocardiography
5. Life expectancy less than one year
6. Cerebro-vascular event within the past 3 months
7. History of mitral/tricuspid endocarditis within the last 12 months
8. Patient has untreated significant left sided valvular heart disease which requires treatment (e.g. mitral regurgitation or stenosis, and aortic regurgitation or stenosis)
9. Documented primary coagulopathy or platelet disorder, including thrombocytopenia (absolute platelet count <90k)
10. Documented evidence of significant renal dysfunction (serum creatinine > 3.0mg/dl) or on any form of dialysis at time of screening within the last 4 weeks
11. Contraindication or known allergy to device's components, anti-coagulation therapy with vitamin K antagonists or contrast media that cannot be adequately pre-treated
12. Patients unsuitable for implantation because of thrombosis of the lower venous system or vena cava filter
13. Evidence of an acute myocardial infarction (AMI) ≤ 1 month (30 days)
14. Liver cirrhosis Child C
15. Female patient of child-bearing potential
16. Currently participating in another study of an investigational drug or device that would directly impact the treatment or outcome of the current study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe, massive or torrential tricuspid regurgitation (TR) undergoing TricValve implantation from multiple Italian and European centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The composite of all-cause mortality and HF rehospitalization at 6-month follow-up | 6-month follow-up
  The composite of all-cause mortality and HF rehospitalization at 6-month follow-up

SECONDARY OUTCOMES:
The composite of all-cause mortality and HF rehospitalization at 1-year follow-up | 1-year follow-up
  The composite of all-cause mortality and HF rehospitalization at 1-year follow-up
Cardiovascular mortality at 1-year follow-up | 1-year follow-up
  Cardiovascular mortality at 1-year follow-up
Number of HF rehospitalizations at 1-year follow-up | 1-year follow-up
  Number of HF rehospitalizations at 1-year follow-up
Number of unscheduled cardiology consultations resulting in changes in medical therapy at 6- month follow-up. | 6- month follow-up
  Number of unscheduled cardiology consultations resulting in changes in medical therapy at 6- month follow-up.
Change in New York Hearts Association (NYHA) functional class and change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score at 6-month and 1-year follow-up. | 6- month follow-up
  Change in New York Hearts Association (NYHA) functional class and change in Kansas City Cardiomyopathy Questionnaire (KCCQ) score at 6-month and 1-year follow-up.
Change in the dose of loop diuretics (in mg/day) at 6-month follow-up | 6- month follow-up.
  Change in the dose of loop diuretics (in mg/day) at 6-month follow-up
Progression of kidney disease, defined as the composite of end-stage kidney disease, a decrease in eGFR to <10 ml/min/1.73 m2, a decrease in eGFR ≥40% from baseline, and death from renal causes at 6-month follow-up. | 6- month follow-up.
  Progression of kidney disease, defined as the composite of end-stage kidney disease, a decrease in eGFR to <10 ml/min/1.73 m2, a decrease in eGFR ≥40% from baseline, and death from renal causes at 6-month follow-up.
Change in 6MWD and in peak oxygen uptake (VO2) at 6-month follow-up. | 6- month follow-up.
  Change in 6MWD and in peak oxygen uptake (VO2) at 6-month follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero Universitaria Pisana, Pisa, Italy